CLINICAL TRIAL: NCT03078569
Title: Transdermal Testosterone for Poor Responders Undergoing IVF
Brief Title: Transdermal Testosterone for Poor Responder Patients Undergoing Controlled Ovarian Stimulation Prior to IVF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, amir shalev, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wolfson testosterone 1
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Infertility, Female
Keywords: Poor responders
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- testosterone gel (Experimental): testosterone gel treatment group
  Interventions: Drug: Testosterone gel
- Control group (No Intervention): without testosterone treatment

INTERVENTIONS:
Drug: Testosterone gel — treatment with testosterone gel
  Other Names: testomax
  Arms: testosterone gel

SUMMARY:
This study evaluates the efficacy of pre- IVF treatment with transdermal testosterone to enhance ovarian response in poor responders.

a randomized controlled trial with two groups, treatment group with transdermal testosterone before IVF treatment and a control group with no treatment.

DETAILED DESCRIPTION:
One of the major challenges of Assisted reproduction technology is treating women with low ovarian response,those women achieve very poor pregnancy rate with IVF.

in recent years there is a focus

ELIGIBILITY:
Inclusion Criteria:

* infertility patients undergoing ART regular menses normal function of thyroid, liver and kidney normal BMI (19.3-28.9) without use of any fertility drugs in the previous two months

Exclusion Criteria:

* patients with recurrent implantations failure (3 cycles and more) previous ovarian surgery uncontrolled medical illness severe endometriosis (stage 3-4) contraindication for testosterone use

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only women under IVF treatment
Enrollment: 30 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
number of retrieved oocytes | 2 year
  number of oocytes

SECONDARY OUTCOMES:
number of clinical pregnancies | 2.5 years
  number of pregnancies with fetal cardiac activity

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson MC, Holon, Israel

IPD SHARING:
Plan to Share IPD: No